CLINICAL TRIAL: NCT04190914
Title: Clinical and Radiographic Evaluation of Triple Antibiotic Paste and Calcium Hydroxide With Iodoform as Intra-canal Medications in Regenerative Treatment of Necrotic Primary Teeth Randomized Clinical Trial
Brief Title: Different Treatment Modality in Necrotic Primary Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: dina darwish (Other)
Responsible Party: Sponsor-Investigator, dina darwish, assistant lecture, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PED18-4D
Record Dates: First submitted 2019-12-05; First posted 2019-12-09 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-11

CONDITIONS: Primary Teeth; Dental Pulp Regeneration
Keywords: triple antibiotic paste

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: participant and outcomes assessor will be blind to which group they belong or assess respectively
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- necrotic primary molar treated with pulpectomy followed by SSC (Active Comparator): control group treated by pulpectomy under rubber dam isolation access cavity will be prepared by a round bur then filling and irrigation will be performed and the tooth will be restored with a temporary filling. After one week all signs and symptoms will be assessed in case of absence of signs and symptoms the tooth will be restored with zin oxide and eugenol and SSC
  Interventions: Other: pulp regeneration for necrotic primary teeth
- necrotic primary molar treated with regeneration using triple (Experimental): under rubber dam isolation access cavity will be prepared by a round bur then minimal filling and irrigation will be performed then triple antibiotic paste will be inserted into the canals and the tooth will be restored by a glass ionomer (GI) as a temporary filling. After2-4 weeks all signs and symptoms will be assessed in case of absence of signs and symptoms an endodontic file will be used to induce bleeding from the periapical area after hemostasis mineral trioxide aggregate will be applied followed by SSC
  Interventions: Other: pulp regeneration for necrotic primary teeth
- necrotic primary molar treated with regeneration using metape (Experimental): under rubber dam isolation access cavity will be prepared by a round bur then minimal filling and irrigation will be performed then calcium hydroxide with iodoform (metapex) will be inserted into the canals and the tooth will be restored by a glass ionomer (GI) as a temporary filling. After 2-4 weeks all signs and symptoms will be assessed in case of absence of signs and symptoms an endodontic file will be used to induce bleeding from the periapical area after hemostasis mineral trioxide aggregate will be applied followed by SSC
  Interventions: Other: pulp regeneration for necrotic primary teeth

INTERVENTIONS:
Other: pulp regeneration for necrotic primary teeth — a pulp regeneration procedure will be applied for necrotic primary teeth with different intracanal medication compared to conventional pulpectomy used in treatment for necrotic primary teeth
  Other Names: different treatment options for necrotic primary teeth

SUMMARY:
Necrotic primary molars in preschool children will be treated with the regeneration concept to provide a healthy biological environment within the root canal system and regression in clinical signs and symptoms which are the primary outcomes of regeneration treatment.

DETAILED DESCRIPTION:
A convenient sample of preschool children have a necrotic primary second molar randomly allocated to one of the 3 study groups which are: group A (control) treated by the conventional treatment ( pulpectomy followed by stainless steel crown SSC), group B: treated by regeneration using triple antibiotic paste followed by SSC), group 3:(treated by regeneration using calcium hydroxide with iodoform(metapex) followed by SSC.

the 3 groups were evaluated at baseline, 6 months and 12 months for clinical and radiographic success.

ELIGIBILITY:
Inclusion Criteria:

* A child with one or more necrotic primary teeth
* Presence of abscess/fistula
* Sensitivity to percussion
* Presence of maximum grade 2 mobility ( Not more than 1 mm)
* Increases of the dental lamina dura
* cooperative patients

Exclusion Criteria:

* Medically compromised children
* Patient allergic to any of the used materials
* Presence of pathologic root resorption (internal-external) or more than 1/3 of the apical root.
* Presence of vitality in the canals
* Presence of grade 3 mobility
* Non-restorable teeth

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2020-02-07 (Actual); Primary Completion 2021-09-07 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
number of patients treated in the 3 groups and have a clinical success according to the checklist absence of pain, pain on percussion, mobility, clinical abscess or fistula | 12 months
  the blind outcome assessor will evaluate the clinical success at 6 and 12 years
number of patients treated in the 3 groups and have a radio graphic success according to the checklist absence of radiolucency, internal or external root resorption | 12 months
  the blind outcome assessor will evaluate the radio graphic success at 6 and 12 years

CONTACTS AND LOCATIONS:
Overall Officials: Dina D Abd-Elmoneam, masters, Principal Investigator — Ain Shams University
Locations (1):
- Faculty of Dentistry- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abdelmoneim DD, Abdelaziz AM, Allam GG, Badran AS. A 1-year Clinical and Radiographic Assessment of Regenerative Endodontic Therapy for Necrotic Primary Molars: A Randomized controlled Trial. Int J Clin Pediatr Dent. 2023 Mar-Apr;16(2):295-301. doi: 10.5005/jp-journals-10005-2536. PMID 37519971